CLINICAL TRIAL: NCT02831088
Title: A Phase II, Double-blind, Randomized, Placebo-controlled, Multi-center Study to Assess Efficacy and Safety of Neu2000KWL in Patients With Acute Ischemic Stroke Receiving Endovascular Therapy
Brief Title: Safety and Optimal Neuroprotection of neu2000 in Ischemic Stroke With Endovascular reCanalizion (SONIC)
Acronym: SONIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GNT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Neu2000KWL-P01
Record Dates: First submitted 2016-07-03; First posted 2016-07-13 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2016-12

CONDITIONS: Ischemic Stroke
Keywords: Neu2000KWL; Neuroprotection; endovascular therapy; glutamate; free radical
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neu2000KWL High-dose group (Experimental)
  Interventions: Drug: Neu2000KWL High-does group
- Neu2000KWL Low-dose group (Experimental)
  Interventions: Drug: Neu2000KWL Low-does group
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neu2000KWL High-does group — 1st infusion of 750mg in patients receiving endovascular therapy within 8 hours following ischemic stroke onset followed by 9 consecutive infusions of 500 mg at intervals of 12 hours
  Other Names: Neu2000KWL is produced by GNT Pharma Pharmaceutical company
  Arms: Neu2000KWL High-dose group
Drug: Neu2000KWL Low-does group — 1st infusion of 500mg in patients receiving endovascular therapy within 8 hours following ischemic stroke onset followed by 9 consecutive infusions of 250 mg at intervals of 12 hours
  Other Names: Neu2000KWL is produced by GNT Pharma Pharmaceutical company
  Arms: Neu2000KWL Low-dose group
Drug: Placebo — 1st infusion of the same volume of saline in patients receiving endovascular therapy within 8 hours following ischemic stroke onset followed by 9 consecutive infusions of same volume of saline at intervals of 12 hours
  Arms: Placebo

SUMMARY:
Efficacy and safety of Neu2000, a multi-target drug designed to prevent both NMDA receptor-mediated excitotoxicity and free radical toxicity, will be investigated in acute ischemic stroke patients receiving endovascular treatment to remove clot within 8 hours following stroke onset. Neu2000KWL will be administered before endovascular treatment.

DETAILED DESCRIPTION:
Neu2000 was designed as a multi-target neuroprotectant preventing both the NMDA receptor, a Ca2+-permeable glutamate receptor, and free radicals, two major routes of brain cell death in stroke. Neu2000 is a moderate NR2B-selective NMDA receptor antagonist and spin trapping molecule (=free radical scavenger or antioxidant). Therapeutic potential of Neu2000 has been well demonstrated in four animal models of stroke with better efficacy and therapeutic time windows than either NMDA receptor antagonist or anti-oxidant advanced to clinical trials. In human phase I studies of 165 healthy subjects conducted in the United States and China, Neu2000KWL showed promising safety profiles without any serious adverse events up to a single intravenous infusion of 6000 mg that is far beyond the therapeutic target dose determined in animal models of transient ischemic stroke. Very recently, acute endovascular recanalization therapy has been introduced as the new standard care of care in acute ischemic stroke. The present study is aimed to examine efficacy and safety of Neu2000KWL in acute ischemic stroke patients receiving endovascular thrombectomy within 8 hours of stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥19 years
2. Patients who were presented to hospitals after onset of brain ischemic symptoms from the base of last normal state and can start Endovascular therapy in accordance with standard practice guidelines within 8 hours after the symptom onset.
3. NIHSS scores on screening time point (admission) ≥ 8 points
4. Patients whose activity is possible without the help of others in the gen-eral condition one day before the ischemic stroke onset. and whose Barthel index scores exceed 90 points
5. Patients whose brain CT and CT angiography imaging confirmed acute ischemic stroke and symptomatic intracranial occlusion at screening and whose occlusion site considered the cause of acute ischemic stroke meets the following conditions:

   ① Carotid T or L type occlusion

   ② M1 MCA

   ③ M1-MCA equivalent (two or more M2-MCAs) However, anterior temporal artery is not regarded M2
6. Patients with ASPECTS on Brain CT without early imaging hyper-enhancement ≥ 6
7. Patients who spontaneously submitted a written informed consent to participation on this clinical study

Exclusion Criteria:

1. a medical history of hypersensitivity against aspirin (salicylates), sulfasalazine or (5-ASA) at screening.
2. Patients who meets the exclusion criteria on imaging in intra-arterial re-canalization therapy ① CTA

   Patients whose imaging shows that the site of occlusion considered the cause of acute ischemic stroke meets the following conditions:

   A. MCA + PCA or MCA+ACA occlusion in Carotid T/L B. occlusion of a bilateral large artery C. simultaneous infiltration of anterior and posterior circulation

   ② absence of the collateral circulation corresponding to one of the followings: A. On CT angiography (MIP-CTA) imaging, absence or minimal collateral circulation at ≥50% of MCA territories, compared with pial filling of contralateral side of the lesion.
3. Patients whose heart diseases corresponding to following conditions were confirmed at screening:

   ① Patients who were diagnosed with myocardial infarction within 6 months at screening

   ② Patients who had severe arrhythmia evoking clinical symptoms (respiratory difficulties, tachycardia etc.) within 6 months at screening.

   Patients whose ECG measured at the stable state at emergency room confirmed the following results:

   A. pulse rate < 50 or >120 beats per minute B. 2nd or 3rd degree AV block is confirmed. C. congenital or acquired QT syndrome is confirmed D. ventricular pre-excitation syndrome is confirmed
4. Patients who were diagnosed with heart failure ≥ class II according to "heart failure classification by NYHA (New York Heart Association)" before screening.

   "heart failure classification by NYHA (New York Heart Association)" Class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities.

   Class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion.

   Class III: patients with marked limitation of activity; they are comfortable only at rest.

   Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on.
5. Patients who have contraindication to contrast media for brain imaging
6. Patients who are receiving renal replacement therapy such as dialysis, due to acute or chronic renal failure, nephropathy, etc. at screening.
7. Patients who were diagnosed with cancer or received cancer therapy within 6 months at screening or have recurrent or transitional cancer
8. Patients who show high body temperature of 38℃ or more or who need antibiotic therapy due to medical opinion of infectious diseases at screening.
9. Patients who take pharmacotherapy due to liver diseases such as hepatitis, liver cirrhosis etc. at screening.
10. Patients who are pregnant or lactating. However, in case of a woman of child-bearing potential, only patients whose non-pregnancy was confirmed can participate in this clinical study.
11. Patients who participated in other clinical studies within past 3 months at the screening time as a base. However, in case of participation in an observatory study without medication, the patients can participate in this clinical study.
12. Patients who were determined unsuitable for participation in this clinical study due to other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportional Ratios of study subjects with mRS 0-2 scores at 12 weeks after Neu2000KWL treatment | 12weeks
Occurrence rate of cerebral hemorrhagic transformation occurring within 48 hours based on parenchymal hematoma (PH) criteria by ECASS (European Co-operative Acute Stroke Study)-I and II | 12weeks

SECONDARY OUTCOMES:
Distribution changes of mRS scores at 1, 4 and 12 weeks vs baseline (shift analysis) | 1week, 4weeks, 12weeks
Ratios of NIHSS 0-2 scores at 1, 4 and 12 weeks vs baseline | 1week, 4weeks, 12weeks
Ratios of Barthel index >90 (≥ 95) at 1, 4 and 12 weeks vs baseline | 1week, 4weeks, 12weeks
Occurrence rate of cerebral hemorrhagic transformation occurring within Day 4 or Day 5 (Day of the last treatment of the study drug) | 4-5days
  based on parenchymal hematoma (PH) criteria by ECASS (European Co-operative Acute Stroke Study)-I and II
Occurrence rate of symptomatic intracranial hemorrhage (SICH) described and defined by this study protocol occurring within Day 4 or Day 5 (Day of the last treatment of the study drug) | 4-5days
  It is defined as SICH of intracranial hemorrhage by brain imaging is confirmed and any one of the following conditions is accompanied:
  A. in case that NIHSS scores become worse 2 points or more B. in case that NIHSS scores become worse 1 point or more, accompanying decreased consciousness C. in case that neurological deficits persist 24 hours or more (and), D. in case of recurrence of stroke and progress deterioration, or in case that other medical causes are not related.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Man Hong, MD, PhD, Principal Investigator — Ajou University Medical Centre
Locations (6):
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chosun University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Ajou University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hong JM, Lee JS, Lee YB, Shin DH, Shin DI, Hwang YH, Ahn SH, Kim JG, Sohn SI, Kwon SU, Lee JS, Gwag BJ, Chamorro A, Choi DW; SONIC Investigators. Nelonemdaz for Patients With Acute Ischemic Stroke Undergoing Endovascular Reperfusion Therapy: A Randomized Phase II Trial. Stroke. 2022 Nov;53(11):3250-3259. doi: 10.1161/STROKEAHA.122.039649. Epub 2022 Sep 6. PMID 36065810
- [Derived] Hong JM, Choi MH, Sohn SI, Hwang YH, Ahn SH, Lee YB, Shin DI, Chamorro A, Choi DW; on the behalf of the SONIC investigators. Safety and Optimal Neuroprotection of neu2000 in acute Ischemic stroke with reCanalization: study protocol for a randomized, double-blinded, placebo-controlled, phase-II trial. Trials. 2018 Jul 13;19(1):375. doi: 10.1186/s13063-018-2746-9. PMID 30005644